CLINICAL TRIAL: NCT07362264
Title: An Open, Multicenter, Phase I Clinical Study on the Safety, Efficacy, and Pharmacokinetics of SH006 Injection Combination in Patients With Advanced Solid Tumors
Brief Title: A Study of SH006 Injection Combination Therapy in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHS006-I-02
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH006 (15mg/kg)/SH006 (30mg/kg)+Bevacizumab±Oxaliplatin±Capecitabine Tablet (Experimental)
  Interventions: Drug: SH006

INTERVENTIONS:
Drug: SH006 — The dosage of SH006 is 15 mg/kg Q3W or 30 mg/kg Q3W, with a treatment cycle of 21 days

SUMMARY:
To evaluate the safety and tolerability of the combination therapy of SH006 injection in patients with advanced solid tumors

DETAILED DESCRIPTION:
This is an open-label, multicenter study to evaluate the safety and efficacy of SH006 injection (15 mg/kg/30 mg/kg) in combination with bevacizumab/oxaliplatin/capecitabine in the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is capable of comprehending the informed consent form, voluntarily agrees to participate, and signs the informed consent form.
2. Age 18 to 75 years (inclusive) on the day of signing the informed consent form, both male and female.
3. Patients with advanced solid tumors who have failed at least one line of standard therapy, or for whom no standard therapy exists, or for whom standard therapy is currently not applicable.
4. According to RECIST 1.1 criteria, at least one measurable lesion at baseline (which has not been previously irradiated): accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) (preferred with intravenous contrast) with a long diameter ≥10 mm (except for lymph nodes, whose short axis must be ≥15 mm), and the lesion is suitable for repeated measurement. Lesions previously irradiated can only be considered measurable if there is documented progression in the irradiated lesion or if the lesion persists for more than three months after radiotherapy, and it meets the RECIST 1.1 criteria.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
6. Life expectancy ≥3 months, in the investigator's judgment.
7. Any toxicities from prior anti-tumor therapy have recovered to ≤ Grade 1 as per CTCAE v5.0, with the exception of alopecia, pigmentation, peripheral neuropathy ≤ Grade 2, hypothyroidism managed with hormone replacement, other confirmed chronic adverse events, or toxicities deemed by the investigator to pose no safety risk.
8. Organ function levels must meet the following requirements (no blood transfusion, blood products, or hematopoietic growth factors for correction within 14 days prior to screening):Hematology: Absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥75×10⁹/L, hemoglobin (Hb) ≥90 g/L.

   Liver Function; Albumin (ALB) ≥28 g/L, total bilirubin (TBIL) ≤3× upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5×ULN;Renal Function: Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) >50 mL/min (calculated using the Cockcroft-Gault formula); Coagulation: International normalized ratio (INR) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN, prothrombin time (PT) ≤1.5×ULN; Urinalysis: Urine protein <2+; for subjects with urine protein ≥2+, a 24-hour urine collection must demonstrate a quantitative protein level <1 g/24 hours.
9. For subjects who are hepatitis B surface antigen (HBsAg) positive and/or hepatitis B core antibody (HBcAb) positive, HBV DNA must be <2000 IU/mL. They must continue or initiate anti-HBV therapy (e.g., entecavir, tenofovir disoproxil fumarate) throughout the study. For those not previously on antiviral therapy, it should be initiated within 1 week prior to the first dose or during the study as appropriate;For subjects who are hepatitis C virus antibody (HCV-Ab) positive, HCV RNA must be below the lower limit of detection.
10. Female subjects of childbearing potential must use effective contraception during the trial and for 6 months after the last dose, and have a negative pregnancy test within 7 days prior to treatment initiation; male subjects must practice effective contraception from signing the informed consent until 6 months after the last dose.
11. The subject is capable and willing to comply with the visits, treatment plan, laboratory tests, and other study-related procedures as specified in the study protocol.

Exclusion Criteria:

1. Prior treatment with TIGIT inhibitors (including monoclonal antibodies, bispecific antibodies, or other agents).
2. Administration of any investigational drug within 28 days prior to the first dose in this trial, or concurrent participation in another clinical study, with the following exceptions: participation in an observational, non-interventional clinical study, or being in the follow-up period of an interventional study where treatment ended more than the washout period (28 days after the last dose) ago.
3. Within 3 weeks prior to the first dose in this trial: chemotherapy; or within 4 weeks prior: targeted therapy, endocrine therapy, or immunotherapy, except for the following: mitomycin or nitrosoureas within 6 weeks prior; oral fluoropyrimidines (e.g., S-1, capecitabine) and small-molecule targeted agents within 2 weeks prior. Prior use of traditional Chinese medicine/herbal medicine with anti-cancer activity described in its labeling is permitted, provided it is discontinued before the first dose of the study drug.
4. Radical radiotherapy within 3 months prior to the first dose in this trial. Palliative radiotherapy within 2 weeks prior is allowed if the radiation dose meets local standards for palliative care and covers <30% of the bone marrow area.
5. Major organ surgery (excluding needle biopsy) and/or local therapy within 28 days prior to the first dose, or unhealed wounds, active peptic ulcer, untreated fracture, or planned elective surgery during the study period.
6. Central nervous system (CNS) metastases causing clinical symptoms or requiring therapeutic intervention. Patients with previously treated brain metastases may be eligible if they are asymptomatic, show stable disease on imaging for ≥4 weeks prior to the first dose, and require no corticosteroids or anti-epileptic drugs.
7. History of allogeneic hematopoietic stem cell transplantation or organ transplantation (excluding corneal transplantation).
8. Clinically uncontrollable third-space fluid collection (e.g., pleural effusion, ascites, pericardial effusion) not manageable by drainage or other methods prior to the first dose, as judged by the investigator.
9. Co-infection with HBV and HCV; HIV antibody positive.
10. Requirement for intravenous antibiotics for >7 days within 2 weeks prior to the first dose, systemic infection, or other severe infection.
11. Hemorrhagic symptoms within 2 months prior to the first dose, such as hemoptysis (>2.5 mL of fresh blood) or history of gastrointestinal bleeding, as judged by the investigator to warrant exclusion.
12. Patients with high bleeding risk indicated by endoscopy within 3 months prior to the first dose (e.g., moderate-to-severe red color signs on esophagogastric varices) or other conditions deemed by the investigator to confer bleeding risk (including active gastrointestinal ulcer, Crohn's disease, ulcerative colitis). The investigator will determine the need for endoscopy in other cases.
13. Thrombolytic therapy (e.g., pro-urokinase, reteplase, alteplase, urokinase) or full-dose anticoagulation (e.g., unfractionated heparin) within 14 days prior to the first dose, excluding prophylactic anticoagulants like low-molecular-weight heparin.
14. History of gastrointestinal perforation and/or fistula, abdominal abscess, or intestinal obstruction (including incomplete obstruction requiring parenteral nutrition) within 6 months prior to the first dose.
15. Systemic glucocorticoid (>10 mg/day prednisone equivalent) or other immunosuppressant therapy within 14 days prior to the first dose, except: topical, ocular, intra-articular, intranasal, or inhaled glucocorticoids; short-term prophylactic use (e.g., for contrast media allergy).
16. Severe respiratory disease or interstitial lung disease, as judged by the investigator to warrant exclusion.
17. Anti-tuberculosis treatment within 1 year prior to the first dose.
18. Administration of live (including attenuated) vaccines within 28 days prior to the first dose.
19. Major vascular event (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to the first dose.
20. Severe or uncontrolled systemic disease, including but not limited to: uncontrolled diabetes; ventricular arrhythmia requiring intervention; acute coronary syndrome, congestive heart failure, stroke, or other ≥Grade 3 cardiovascular event within 6 months; NYHA Class ≥II or LVEF <50%; clinically significant QTcF prolongation or arrhythmia risk (baseline QTcF >450 msec for males or >470 msec for females, uncorrectable hypokalemia, long QT syndrome, atrial fibrillation with resting heart rate >100 bpm, or severe valvular disease); clinically uncontrolled hypertension (SBP >150 mmHg and/or DBP >90 mmHg after treatment) as judged by the investigator.
21. History of hypertensive crisis or hypertensive encephalopathy.
22. History or presence of autoimmune disease within 2 years, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's granulomatosis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, Guillain-Barré syndrome, or high risk (e.g., post-transplant immunosuppression). Exceptions: stable type 1 diabetes on fixed-dose insulin; autoimmune hypothyroidism on hormone replacement only; skin conditions not requiring systemic treatment (e.g., eczema, rash covering <10% BSA, psoriasis without ocular symptoms).
23. Prior immunotherapy with ≥Grade 3 irAE or ≥Grade 2 immune-related myocarditis.
24. History or presence of other malignancies, except: (i) cured early-stage malignancies (carcinoma in situ or Stage I), e.g., adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer; (ii) cured second primary cancer with no recurrence within 5 years; (iii) both primaries are expected to benefit from this study, per investigator.
25. Known history of severe hypersensitivity to PD-1/PD-L1 antibodies, VEGF antibodies, or similar macromolecular agents, or severe hypersensitivity (CTCAE v5.0 Grade ≥3) to any component of the study drug.
26. Pregnant or lactating women.
27. Known alcohol and/or drug dependence, or any other condition deemed by the investigator to affect the safety or compliance of the study treatment, including but not limited to psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs) | Days 1-21
Recommended Phase 2 Dose (RP2D) | up to 21 days
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Within 90 days from the first administration to the last administration of the SH006 combination therapy

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 | Every two cycles (each cycle lasting 21 days) until the end of treatment, with an average of 2 years.
Duration of Response (DOR) as Per RECIST v.1.1 | Every two cycles (each cycle lasting 21 days) until the end of treatment, with an average of 2 years.
Progression Free Survival (PFS) as Per RECIST v.1.1 | Every two cycles (each cycle lasting 21 days) until the end of treatment, with an average of 2 years.
DCR as Per RECIST v.1.1 | Every two cycles (each cycle lasting 21 days) until the end of treatment, with an average of 2 years.
overall survival as Per RECIST v.1.1 | Every 2 cycles (each cycle lasting 21 days) until the end of the treatment; Once every 12 weeks until the end of the follow-up, with an average of 2 years.
Maximum Concentration (Cmax) of SH006 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Time of Maximum Concentration (Tmax) of SH006 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Area Under the Curve (AUC) of SH006 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Clearance (CL) of SH006 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
Evaluation of the immunogenicity of SH006 | At pre-defined intervals from initial dose through final study visit (up to 24 months)
  Serum sampling to assess the potential for anti-drug antibody (ADA) formation

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Tianyinshan Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No